CLINICAL TRIAL: NCT00304993
Title: Study of Niacin and Rosiglitazone in Dysmetabolic Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation Research, Florida (Other)
Collaborators: GlaxoSmithKline (Industry); Kos Pharmaceuticals (Industry); Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNARED
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2006-03-21 (Estimated); Status verified 2006-03

CONDITIONS: Metabolic Syndrome X; Insulin Resistance
Keywords: fenofibrate; niacin; rosiglitazone; LDL phenotype pattern B; small, dense LDL; insulin resistance; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Cerebral Palsy | interventions — Fenofibrate; Niacin; Rosiglitazone

INTERVENTIONS:
Drug: fenofibrate
Drug: niacin
Drug: rosiglitazone

SUMMARY:
Lipid abnormalities in people with the Metabolic Syndrome (the Insulin Resistance Syndrome) are characterized by elevations in triglycerides and LDL cholesterol; low levels of HDL cholesterol; and small, dense LDL particles. Statins generally do not change LDL particle size, so often fenofibrate is added. This combination may still not be sufficient. Niacin is a common third drug added to the treatment regimen, but niacin can increase insulin resistance. This study compares niacin as a third drug to rosiglitazone, an insulin sensitizer.

DETAILED DESCRIPTION:
The Metabolic Syndrome is characterized by an atherogenic dyslipidemia consisting of hypertriglyceridemia, modest elevations of LDL cholesterol, low levels of HDL cholesterol, and LDL phenotype pattern B (small, dense LDL particles). Statins are first line therapy, and reduce LDL cholesterol levels without affecting LDL particle size. Fenofibrate addresses the triglycerides, HDL cholesterol levels, and LDL phenotype, so is recommended as second level therapy. The third element is niacin, but for insulin resistant patients, a question has been whether niacin might be exacerbating the underlying pathophysiology of Metabolic Syndrome patients. In SNARED, niacin was compared to the insulin sensitizer rosiglitazone in study subjects already on statin and fenofibrate.

All volunteers participating in SNARED exhibit LDL phenotype pattern B despite statin therapy at the time of recruitment. Comparisons of LDL phenotype at baseline are to be compared to measurements made after 4 months of statin + fenofibrate. If the LDL phenotype converts to pattern A (large LDL particles), this is a study endpoint. Otherwise, study subjcts are randomized to receive statin+fenofibrate+niacin, or statin+fenofibrate+rosiglitazone for six months, at which time lipid phenotype will again be determined..

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years Fasting triglycerides > 100 mg/dL Fasting plasma glucose 110-128 mg/dL Non-pattern A LDL phenotype

Exclusion Criteria:

* Overt diabetes mellitus Current therapy with hypoglycemic agents Secondary causes of dyslipidemia (e.g. HRT, thyroid disease) Serum creatinine > 2.5 mg/dL or nephrotic syndrome AST/ALT > 3X upper limits of normal Known gallbladder disease History of gout or hyperuricemia History of peptic ulcer disease Hypersensitivity or intolerance to any of the study drugs Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-01; Study Completion 2005-02

PRIMARY OUTCOMES:
The effect of treatment on Peak LDL particle size

SECONDARY OUTCOMES:
The effect of treatment on:
traditional lipid parameters (LDL-C, HDL-C, triglycerides)
% of lipids in regions IIIa+IIIb of a gradient gel electrophoresis
LDL phenotype
fasting glucose
Hemoglobin A1c

CONTACTS AND LOCATIONS:
Overall Officials: Michael E McIvor, MD, Principal Investigator — Foundation Research
Locations (1):
- Foundation Research, St. Petersburg, Florida, United States